CLINICAL TRIAL: NCT04423302
Title: Randomized Placebo-controlled Double-blinded Study of the Effect of TOTUM-63 on Glucose and Lipid Homeostasis in Subjects With Dysglycemia
Brief Title: Effect of Totum-63 on Glucose and Lipid Homeostasis in Subjects With Dysglycemia (REVERSE-IT)
Acronym: REVERSE-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valbiotis (Industry)
Collaborators: Biofortis Mérieux NutriSciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PEC16075; 2020-A00604-35 (Other: ID-RCB)
Record Dates: First submitted 2020-05-28; First posted 2020-06-09 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Prediabetic State; Diabetes type2; Dysglycemia
Keywords: Dysglycemia; Prediabetes; Type 2 diabetes; Hyperglycemia; Insulinemia; Diabetes risk; Diet supplement; Plant extracts; Health condition; Hygiene and dietary recommendations; Diet
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2; Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 2 blinded arms (Active 3 intakes per day and Placebo 3 intakes per day) and 1 open arm (Active 2 intakes per day)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TOTUM-63 3 intakes per day (Experimental): Experimental active diet supplement TOTUM-63 taken 3 times per day (blinded arm)
  Interventions: Dietary Supplement: TOTUM-63 3 intakes per day
- Placebo 3 intakes per day (Placebo Comparator): Placebo comparator taken 3 times per day (blinded arm)
  Interventions: Dietary Supplement: Placebo 3 intakes per day
- TOTUM-63 2 intakes per day (Experimental): Experimental active diet supplement TOTUM-63 taken 2 times per day (open arm)
  Interventions: Dietary Supplement: TOTUM-63 2 intakes per day

INTERVENTIONS:
Dietary Supplement: TOTUM-63 3 intakes per day — 5-g dose of TOTUM-63 diet supplement, a mix of 5 plant extracts. Eight capsules per day to consume orally in three intakes (3 in the morning, 2 at lunch and 3 at dinner)
  Other Names: Active product 3 intakes per day
  Arms: TOTUM-63 3 intakes per day
Dietary Supplement: Placebo 3 intakes per day — Placebo. Eight capsules per day to consume orally in three intakes (3 in the morning, 2 at lunch and 3 at dinner)
  Other Names: Comparator product 3 intakes per day
  Arms: Placebo 3 intakes per day
Dietary Supplement: TOTUM-63 2 intakes per day — 5-g dose of TOTUM-63 diet supplement, a mix of 5 plant extracts. Eight capsules per day to consume orally in two intakes (4 in the morning and 4 at dinner)
  Other Names: Active product 2 intakes per day
  Arms: TOTUM-63 2 intakes per day

SUMMARY:
This clinical study aims to assess the efficacy of TOTUM-63, a mix of 5 plant extracts, consumed at the daily regimen of three times per day on glucose and lipid homeostasis in dysglycemic subjects. The hypothesis is that TOTUM-63, consumed 3 times per day, is superior to placebo for decrease of fasting plasma glucose (FPG) concentration after 24 weeks of consumption.

ELIGIBILITY:
Inclusion Criteria:

* I1. From 18 to 70 years (including ranges);
* I2. Dysglycemic, prediabetic or newly diagnosed type 2 diabetes, subject without any clinical symptoms of diabetes (e.g. polyuria, polydipsia, blurred vision…) and not requiring immediate anti-diabetic treatment;
* I3. Body mass index (BMI) between 25 and 40 kg/m² (including ranges);
* I4. Waist circumference > 102 cm for men and > 88 cm for women (-2% margin allowed, respectively ≥ 100 cm and ≥ 86.5 cm);
* I5. Weight stable within ± 5% in the last three months;
* I6. No significant change in food habits or in physical activity in the 3 months before the randomization and agreeing to follow hygiene and dietary (HD) recommendations given during the study;
* I7. For women: Non-menopausal with the same reliable contraception since at least three months before the beginning of the study and agreeing to keep it during the entire duration of the study (hormonal contraception, intra uterine device or surgical intervention) or menopausal with or without hormone replacement therapy (estrogenic replacement therapy begun from less than 3 months excluded);
* I8. Good general and mental health according to the opinion of the investigator: no clinically significant and relevant abnormalities of medical history or physical examination;
* I9. Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form;
* I10. Affiliated with a social security scheme;
* I11. Agreeing to be registered on the volunteers in biomedical research (applicable only for French centers).

At V0 biological analysis, the subjects will be eligible to the study on the following criteria:

* I12. Fasting plasma glucose concentration ≥ 110 mg/dL.

Exclusion Criteria:

* E1. Suffering from a metabolic disorder such as treated diabetes, uncontrolled thyroidal dysfunction or other metabolic disorder needing a dose adjustment in drug intervention according to the professional recommendations;
* E2. Suffering from an uncontrolled arterial hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg);
* E3. With a history of retinopathy, ischemic cardiovascular event, having undergone recent surgical procedure in the past 6 months or in the 9 months to come;
* E4. Suffering from a severe chronic disease (e.g. cancer, HIV, renal failure, hepatic or biliary disorders ongoing, chronic inflammatory digestive disease, arthritis or other chronic respiratory trouble, etc.) or gastrointestinal disorders found to be inconsistent with the conduct of the study by the investigator (e.g. celiac disease);
* E5. Under antidiabetic drug (e.g. biguanides, sulfonylureas, glinides, gliptins, glitazones, gliflozins, α-glucosidase inhibitors, incretins and insulin);
* E6. Under lipid-lowering treatment (e.g. statins, fibrates, ezetimibe, bile acid sequestrants, niacin, etc.) since less than 3 months or modification of the treatment dose since less than 3 months before the randomization. Subject with a stable lipid-lowering treatment since at least three months can be included in the study;
* E7. Under medication which could affect glucose and/or lipid homeostasis parameters or stopped less than 3 months before randomization (e.g. beta 2 agonists like salbutamol, Angiotensin Converting Enzyme (ACE) inhibitors, beta blockers, thiazide diuretics, Selective Serotonin Reuptake Inhibitors (SSRIs), Mono-Amine Oxidase Inhibitors (MAOIs), neuroleptics, long-term corticosteroid systemic drugs, systemic antibodies, androgens, phenytoin, interferons, immunosuppressants, antivirals and antiretrovirals, etc.):

  * Beta 2 agonists like salbutamol, ACE inhibitors, beta blockers, thiazide diuretics, SSRIs, MAOIs are tolerated only if stable since more than 3 months before the randomization and maintained during the whole study;
  * The others drugs (neuroleptics, long-term corticosteroid systemic drugs, systemic antibodies, androgens, phenytoin, interferons, immunosuppressants, antivirals and antiretrovirals, etc.) are not allowed during the study;
* E8. Regular intake of dietary supplements or "health foods", or products rich in plant stanol or sterol (like Pro-Activ® or Danacol® products), rich in long chain omega-3 fatty acids (especially soft gels containing fish oils), or in other substances intended to reduce glycemia (e.g. beta-glucans, konjac, olive leaf extract, berberine, cinnamon, etc.) or stopped less than 3 months before the randomization;
* E9. Under treatment or dietary supplement which could significantly affect parameter(s) followed during the study according to the investigator or stopped in a too short period before the randomization (for example consumed in the month before the randomization);
* E10. With a known or suspected food allergy or intolerance or hypersensitivity to any of the study products' ingredient;
* E11. Consuming more than 3 standard drinks daily of alcoholic beverage for men or 2 standard drinks daily for women or not agreeing to keep his alcohol consumption habits unchanged throughout the study;
* E12. With extreme and/or unbalanced eating habits (e.g. vegetarian, vegan, skipping meals regularly);
* E13. With a personal history of anorexia nervosa, bulimia or significant eating disorders according to the investigator;
* E14. Smoking more than 20 cigarettes daily or not agreeing to keep his smoking habits unchanged throughout the study. The subject should be able not to smoke during the visits (maximum 4 hours);
* E15. Having a lifestyle deemed incompatible with the study according to the investigator including high level of physical activity (defined as more than 10 hours of intense physical activity a week, walking excluded);
* E16. Pregnant (as evidenced by a positive test for β-HCG (Human Chorionic Gonadotropin), i.e. > 5 mUI/mL, realized at V0) or lactating women or intending to become pregnant within 9 months ahead;
* E17. Who made a blood donation in the 3 months before the randomization or intending to make it within 9 months ahead;
* E18. Taking part in another clinical trial or being in the exclusion period of a previous clinical trial;
* E19. Having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros (applicable only for French centers);
* E20. Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision;
* E21. Presenting a psychological or linguistic incapability to sign the informed consent;
* E22. Impossible to contact in case of emergency;
* E23. Any condition assessed by the investigator which could endanger patient safety or the conduct of the study (e.g. device related contraindication for impedancemetry and/or DEXA (Dual-Energy X-ray Absorptiometry) such as pacemaker or electronic implant);

At V0 biological analysis, the subjects will be considered as non-eligible to the study on the following criteria:

* E24. Fasting glucose plasma concentration > 220 mg/dL;
* E25. Fasting blood triglycerides > 2.2 g/L;
* E26. TSH (Thyroid Stimulating Hormone) outside the laboratory normal values;
* E27. Fasting blood LDL (Low Density Lipoprotein) cholesterol > 1.9 g/L or non HDLc (High Density Lipoprotein cholesterol) > 2.2 g/L or any condition requiring a therapeutic dose adjustment during the trial according to the professional recommendations;
* E28. Blood AST (ASpartate amino Transferase), ALT (ALanine amino Transferase) or GGT (Gamma Glutamyl Transpeptidase) > 3 x ULN (Upper Limit of Normal);
* E29. Blood creatinine concentration > 125 μmol/L;
* E30. eGFR estimated Glomerular Filtration Rate, calculated by CKD-EPI (Chronic Kidney Disease-EPIdemiology collaboration) formula) < 60 mL/min/1.73m²;
* E31. Complete blood count (CBC) with hemoglobin < 11 g/dL or leucocytes < 3000 /mm3 or leucocytes > 16000 /mm3 or clinically significant abnormality according to the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 636 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Fasting plasma glucose concentration at V3 with a 3 times a day regimen | V3 (24 weeks of intervention)
  Fasting plasma glucose concentration in mg/dL, TOTUM-63 3/day vs placebo

SECONDARY OUTCOMES:
Evolution of the fasting plasma glucose concentration | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Fasting plasma glucose concentration (in mg/dL), TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of the HbA1c | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  HbA1c (in %), TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of the glycemia at 120 minutes following the 75g glucose intake | V1 (baseline), V2 (12 weeks of intervention), V3 (24 weeks of intervention) and V4 (12 weeks and the end of intervention)
  Glycemia (in mg/dL) at 120 minutes following the 75g glucose intake, TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo (Only for a subgroup of 201 subjects)
Evolution of the fasting insulinemia | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Fasting insulinemia (in mU/L), TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of the HOMA-IR (HOmeostasis Model Assessment of Insulin Resistance) index | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  HOMA-IR index, TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of the HOMA-β (Homeostasis Model Assessment of Beta cells) index | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  HOMA-β index, TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of the QUICKY (QUantitative Insulin sensitivity ChecK Index) index | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  QUICKY index, TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of the fasting blood concentrations of triglycerides | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Triglycerides (in g/L), TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of the fasting blood concentrations of total cholesterol | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Total cholesterol (in g/L), TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of the fasting blood concentrations of HDL cholesterol | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  HDL cholesterol (in g/L), TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of the fasting blood concentrations of non-HDL cholesterol | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  non-HDL cholesterol (in g/L), TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of the fasting blood concentrations of LDL cholesterol | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  LDL cholesterol (in g/L), TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of the fasting blood concentrations of free fatty acids | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Free fatty acids (in g/L), TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of atherogenic index | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Atherogenic index, TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of atherogenic coefficient | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Atherogenic coefficient, TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of Cardiac risk ratio 1 | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Cardiac risk ratio 1, TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of cardiac risk ratio 2 | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Cardiac risk ratio 2, TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of the fasting blood concentrations of hsCRP | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  hsCRP (in mg/L), TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of the body weight | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Body weight (in kg), TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of the waist circumference | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Waist circumference (in cm), TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of the hip circumference | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Hip circumference (in cm), TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of the waist to hip ratio | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Waist to hip ratio, TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Evolution of the body composition assessed by impedancemeter | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Fat mass (in % and kg), lean mass (in % and kg), total body water (in % and kg), TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Delay of occurence of pharmacological treatment requirement for type 2 diabetes from V1 | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Delay between V1 and the date at which the investigator will decide to withdraw the subject from the study because he needs a pharmacological treatment to treat his diabetes, TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo
Proportion of subjects having an improvement or a deterioration of their glycemic status from V1 | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Glycemic status will be defined at each visit by the FPG value, 3 different categories Type 2 diabetes/prediabetic/normal. Proportion of subjects changing from category during the study will be assessed during the study (improvement of the glycemic status or deterioration), TOTUM-63 3/day vs placebo, TOTUM-63 2/day vs placebo and TOTUM-63 3/day pooled with TOTUM-63 2/day vs placebo

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle METREAU, MD, Principal Investigator — Biofortis Mérieux NutriSciences
Locations (52):
- Bulgaria (8):
  - MHAT-Botevgrad EOOD, Botevgrad, Botevgrad
  - MHAT Sveta Karidad, First department of Internal Diseases, Plovdiv
  - Ambulatory for IPSOC in Endocrynology and Metabolic Diseases ENDO MED-CONSULT EOOD, Plovdiv
  - Diagnostic-consultative center 7 EOOD, Plovdiv, Plovdiv
  - Diagnostic Consultative Center "ALEXANDROVSKA", Sofia
  - University Multiprofile Hospital for active treatment "Alexandrovska" EAD Clinic of Endocrinology and metabolic diseases, Sofia
  - 4th Multiprofile Hospital for active treatment - EAD, Internal Diseases Departement, Sofia
  - Diagnostic Consultative Center, Sofia
- France (14):
  - CHU Amiens, Amiens
  - CH Arras, Arras
  - CIC Clermont Ferrand, Clermont-Ferrand
  - CEN Nutriment, Dijon
  - Eurofins Optimed, Gières
  - CHU Grenoble, Grenoble
  - Institut Pasteur de Lille, Lille
  - CHU Lille, Lille
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - Unité d'Investigation Clinique Biofortis Mérieux NutriSciences, Paris
  - Unité de Recherche Clinique en Immunologie Lyon Sud, Pierre-Bénite
  - CHU Rouen, Rouen
  - Biofortis Mérieux NutriSciences, Saint-Herblain
- Germany (11):
  - Analyze & Realize, Berlin
  - Klinische Forschung Dresden, Dresden
  - Medizentrum Essen Borbeck, Essen
  - Biotesys, Esslingen am Neckar
  - Klinische Forschung Hamburg, Hamburg
  - Klinische Forschung Hannover-Mitte, Hanover
  - Klinische Forschung Karlsruhe, Karlsruhe
  - Gemeinschaftspraxis Dr. Med C. Klein/J Minnich, Künzing
  - Zentrum fur Klinische Studien, Sankt Ingbert
  - Klinische Forschung Schwerin, Schwerin
  - Zentrum für Klinische Ernährung Stuttgart, Stuttgart
- Hungary (8):
  - Drug Resesarch Center (DRC), Balatonfüred
  - Trial Pharma Ltd, Békéscsaba
  - ClinExpert Medical Center, Budapest
  - Agria - Study Ltd, Eger
  - Trial Pharma Ltd, Győr
  - Trial Pharma Ltd, Gyula
  - Clinical Research Unit (CRU), Miskolc
  - Trial Pharma Ltd, Orosháza
- Italy (4):
  - Azienda Ospedaliera Universitaria "Mater Domini", Catanzaro
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Universitaria Policlinico "Paolo Giaccone", Palermo
  - Policlinico Umberto I, Roma
- Poland (3):
  - Vitamed, Bydgoszcz
  - Grupowa Praktyka Lekarska s.c, Katowice
  - Centrum Medyczne Linden, Krakow
- Romania (4):
  - Sana Monitoring, Bucharest
  - Spitalul Municipal Caracal, Caracal
  - Ames Research Cente, Călăraşi
  - Clintrial Medical Center, Reșca

IPD SHARING:
Plan to Share IPD: No